CLINICAL TRIAL: NCT01661257
Title: Expression of T-cell Immunoglobulin- and Mucin-domain-containing Molecule 3 (TIM-3)and Correlation With Disease Activity in Pediatric Crohn's Disease With Anti TNF-α Therapy
Brief Title: Expression of TIM-3 and Correlation With Disease Activity in Pediatric Crohn's Disease With Anti TNF-α Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, YonHo Choe, Pediatrics, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-10-038-002
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Infliximab; T-cell immunoglobulin- and mucin-domain-containing molecule 3 (TIM-3)
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TIM-3 (Experimental): T-cell immunoglobulin- and mucin-domain-containing molecule 3 (TIM-3) is a novel transmembrane protein that is involved in the regulation of Th1-cell-mediated immunity.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab
  Other Names: Remicade

SUMMARY:
This study investigated the expression of T-cell immunoglobulin- and mucin-domain-containing molecule 3 (TIM-3) in the colonic mucosa and/or the peripheral blood of children with Crohn's disease during anti TNF-α (infliximab) therapy.

DETAILED DESCRIPTION:
The immunoregulatory effects of TIM-3 on patients with Crohn's disease according to the treatment have not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* •Pediatric patients who were diagnosed with severe Crohn's disease who require infliximab treatment

  * confirmed diagnostic of Crohn's disease in clinical, endoscopic and histological findings

Exclusion Criteria:

* •patients who has proven to have infliximab antibody

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Expression of TIM-3 and Correlation With Disease Activity in Pediatric Crohn's Disease with anti TNF-α Therapy | 1-year treatment period
  Disease Activity Index (PCDAI) scores, Peripheral blood for TIM-3 mRNA expression

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea